CLINICAL TRIAL: NCT03716011
Title: A Large, Prospective, Randomized, Multicenter Clinical Study Evaluating the Safety and Efficacy of the Post-marketing Drug-eluting Stent System (Rapamycin) - the EXCROSSAL Stent in CAD Patients With 3-month DAPT or 12-month DAPT
Brief Title: A Postmarket Clinical Trial for EXCROSSAL Stent in CAD Patients With 3-month DAPT or 12-month DAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DREAM-201810
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: the EXCROSSAL stent in CAD patients with 3-month DAPT or 12-month DAPT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAPT 3M or DAPT 12M (Other): After stent implantation in DAPT 3M or DAPT 12M
  Interventions: Device: EXCROSSAL

INTERVENTIONS:
Device: EXCROSSAL — a Second Generation Biodegradable Polymer Sirolimus-Eluting Stent

SUMMARY:
1. Prospective, randomized, multicenter clinical study
2. This is a post-marketing clinical study to evaluate whether it will affect the safety event when it is used in different treatment ways. Adopting non - inferiority design, 2700 cases were enrolled.
3. EDC system (eCRF electronic data collection system)
4. Follow-up points: 30 days,3 months, 12 months, 24 months, 36 months, 48 months and 60 months after the operation;

DETAILED DESCRIPTION:
1. Subjects are eligible for coronary intervention
2. The lesion needs to be pre-expanded or special circumstances should be carefully considered according to the clinical manifestations
3. The selection of target vessel is based on the criteria of a diameter between 2.25mm and 4.0mm
4. If a stent needs to be placed at the target vessel, it is recommended that there be at least 2mm overlap between the stents; if the stent expansion is not sufficient, post-dilatation treatment is required.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years;
2. De novo coronary artery primary lesions;
3. Stable angina pectoris;
4. Patients with coronary artery disease with similar symptoms of myocardial ischemia or angina;
5. Suitable for PCI indication and suitable for the implant of EXCROSSAL stents.
6. Able to understand the purpose of the study, voluntarily participate and sign the informed consent form, and willing to accept the clinical follow-up; Imaging criteria The target lesion length≤ 60mm；Visual reference diameter of the vessel is 2.25-4.0mm;

Exclusion Criteria:

1. Patients with acute myocardial infarction (AMI) within 7 days; Non-ST elevated ACS patients
2. those who implanted any stent before;
3. Left ventricular ejection score(LVEF) 30 %
4. Patients with bleeding tendency or anticoagulation treatment contraindications and/or PCI contraindications or coagulopathy;
5. There are other diseases such as cancer, malignant tumor, congestive heart failure, organ transplant, or candidate) or has a history of abuse (alcohol, cocaine, heroin, etc.), plan adherence is poor, or the life expectancy of less than 1 year;
6. It is estimated that elective surgery patients within 12 months;
7. Other coronary lesions requiring staged intervention;
8. If there are branches of blood vessels that need to be treated, the diameter of blood vessels ≥ 2.5 mm;
9. The subject's compliance or the researcher's judgment was not suitable for the participants in the study;
10. Pregnant or lactating persons; Imaging criteria

1. Left main disease, transplanted vessel lesions, stent restenosis; 2. The balloon cannot be predilated or/or the severe calcification lesion of rotatory failure; 3. The distortion of the stent is difficult to pass;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2018-12-20 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure at 12-Month | 12-month
  The target lesion failure (TLF) rate at 12 months after operation involves cardiac death, target-vessel myocardial infarction, and clinical-symptom driven target vessel revascularization.

SECONDARY OUTCOMES:
MACE rate | 1-month,3-month,6-month, 12-month, 24-month, 36-month, 48-month and 60-month.
  Incidence of major adverse cardiac events (MACE) at different follow-up points of 1-month,3-month,6-month,12-month,24-month,36-month,48-month,60-montjh.
  2. Stent implantation success rate (covering the device success, the lesion success and the clinical success); 3. Target lesion failure (TLF) at 30 days,3 months, 12 months, 24 months, 36 months, 48 months and 60 months after the operation; 4. Subject-related cardio-clinical composite end points at the follow-up points: 30 days,3 months, 12 months, 24 months, 36 months, 48 months and 60 months after the operation, covering all-cause mortality, all myocardial infarctions and any revascularization; 5. The incidence of ARC-defined stent thrombosis events (defined, probable and non-excludable stent thrombosis in early, late, and delayed stages);
Device success rates , lesion success rates , clinical success rates | 1-month,3-month,6-month, 12-month, 24-month, 36-month, 48-month and 60-month.
  The success of the instrument refers to the degree of stenosis in the final bracket after the instrument was implanted. Lt; 30 %(visual), TIMI level 3 blood flow, and no residual stenosis and thrombus.
  The success of the lesion refers to the degree of ultimate diameter stenosis of the target lesion after the application of any interventional treatment. 50 %(visual), TIMI level 3 blood flow, and no residual stenosis and thrombus.
  The success of surgery refers to the absence of major cardiac adverse events caused by ischemia during the patient's hospitalization(up to 7 days after surgery) based on the success of the lesion.
Definite and probable stent thrombosis | 1-month,3-month, 12-month, 24-month, 36-month, 48-month and 60-month.
  According to ARC definition

CONTACTS AND LOCATIONS:
Overall Officials: Hao M Lu, Ph.D, Study Director — Zhongshan hospital of ShangHai FuDan University
Locations (1):
- JW Medical System, Beijing, Beijing Municipality, China